CLINICAL TRIAL: NCT01935622
Title: Phase II Study of Safety and Efficacy of Doxycycline in Patients With Non-Ischemic Cardiomyopathy
Brief Title: Safety and Efficacy of Doxycycline in Patients With Non-Ischemic Cardiomyopathy
Acronym: DOXY-HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End of funding
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCU HM14393
Record Dates: First submitted 2013-08-23; First posted 2013-09-05 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Non-ischemic Cardiomyopathy; Systolic Heart Failure (NYHA II-III)
Keywords: heart failure; non-ischemic cardiomyopathy
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Doxycycline 100 mg (Experimental): Doxycycline 100 mg twice daily for 14 days
  Interventions: Drug: Doxycycline
- Doxycycline 20 mg (Experimental): Doxycycline 20 mg twice daily for 14 days
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 1 tablet every 12 hours for 14 days
  Arms: Doxycycline 100 mg; Doxycycline 20 mg
Drug: placebo — Placebo 1 tablet every 12 hours for 14 days
  Arms: Placebo

SUMMARY:
Non-ischemic cardiomyopathy and heart failure are highly influenced by the presence of systemic inflammation.

Doxycycline is a FDA-approved drug to treat bacterial infections which also shows powerful anti-inflammatory effects.

In this study we plan to determine the effects of Doxycycline in patients with stable heart failure and non-ischemic cardiomyopathy on peak of aerobic exercise capacity (peak V02) and ventilator efficiency measured with a cardiopulmonary test.

DETAILED DESCRIPTION:
In this study of Safety and Efficacy of Doxycycline in Patients with Non-Ischemic Cardiomyopathy Population, we will enroll 24 patients with a clinical diagnosis of heart failure and non-ischemic cardiomyopathy (recent imaging study documenting LV ejection fraction <50%, and no history of coronary or ischemic heart disease) in a single-center, randomized, double-blinded, placebo-controlled clinical trial with allocation 1:1:1 to Doxycycline 100 mg twice daily or Doxycycline 20 mg twice daily or Placebo for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non-ischemic cardiomyopathy (LVEF<40%)
* Heart failure NYHA II-III

Exclusion Criteria:

* Age <18
* Recent changes (previous 3 months) in HF maintenance medications (beta-blockers, angiotensin converting enzyme [ACE] inhibitors, aldosterone antagonists, vasodilators, cardiac glycosides, diuretics)
* Hospitalization for worsening HF or acute decompensated HF within the previous 12 months
* History of coronary or ischemic heart disease
* Anticipated need for cardiac resynchronization therapy (CRT) or automated-implantable cardioverter defibrillator (AICD) or coronary revascularization or cardiac surgery
* Angina or electrocardiograph (ECG) changes that limit maximum exertion during cardiopulmonary exercise testing
* Active infection including chronic infection
* Active cancer (or prior diagnosis of cancer within the past 10 years)
* Recent (<14 days) use of anti-inflammatory drugs (not including NSAIDs), Chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus), malignancy, or any comorbidity limiting survival or ability to complete the study
* Pregnancy
* Inability to give informed consent
* Other conditions limiting completion of cardiopulmonary exercise test or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline 100 mg: Doxycycline 100 mg twice daily for 14 days
  Doxycycline
- Doxycycline 20 mg: Doxycycline 20 mg twice daily for 14 days
  Doxycycline
Period: Overall Study
Arm/Group | Doxycycline 100 mg | Doxycycline 20 mg | Placebo
Started | 3 | 3 | 4
Completed | 1 | 1 | 4
Not Completed | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: (No data analysis conducted. Insufficient enrollment)
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline 100 mg | Doxycycline 20 mg | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Continuous [Median (Full Range); unit: years] | 52 [48 to 55] | 58 [55 to 59] | 54 [49 to 60] | 54 [48 to 60]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 10
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2
  Male | 3 | 3 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Peak Aerobic Exercise Capacity
Description: Interval change in peak VO2 measured at cardiopulmonary test
Time Frame: 14 days
Measure: Median (Inter-Quartile Range)
Arm/Group | Doxycycline 100 mg | Doxycycline 20 mg | Placebo
Number analyzed (Participants) | 3 | 3 | 4
Value | NA [NA to NA] — (No data analysis conducted. Insufficient enrollment) | NA [NA to NA] — (No data analysis conducted. Insufficient enrollment) | NA [NA to NA] — (No data analysis conducted. Insufficient enrollment)

ADVERSE EVENTS:
Arm/Group | Doxycycline 100 mg | Doxycycline 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline 100 mg (N=3) | Doxycycline 20 mg (N=3) | Placebo (N=4)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
(No data analysis conducted. Insufficient enrollment)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No